CLINICAL TRIAL: NCT01083927
Title: Rotational Narrow Strip Versus Full Conjunctival Graft in Pterygium Excision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Dr Lo Sheau Kang, University Malaya Eye Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMERC003
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Pterygium
Keywords: Pterygium
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rotational Narrow Strip Graft (Active Comparator): Technique of surgery
  Interventions: Procedure: Rotational Narrow Strip Conjunctival Graft
- Full Graft (Active Comparator): Surgical technique
  Interventions: Procedure: Full Conjunctival Graft

INTERVENTIONS:
Procedure: Rotational Narrow Strip Conjunctival Graft — Surgical technique
  Arms: Rotational Narrow Strip Graft
Procedure: Full Conjunctival Graft — Surgical technique
  Arms: Full Graft

SUMMARY:
To compare the efficacy of rotational narrow strip conjunctival graft to full conjunctival graft in primary pterygium excision. Risk analysis of factors that may affects the recurrence rate.

DETAILED DESCRIPTION:
Pterygium is a raised, wing-shaped growth of fibrovascular tissue that extends horizontally from the bulbar conjunctiva, crossing the limbus, and onto the cornea. It is a common ocular surface disease in Malaysia.

Pterygium can cause chronic ocular irritation, redness, tearing, visual impairment and poor cosmesis. Treatment of symptomatic pterygium remains surgical. Surgery should achieve low recurrence rate and acceptable cosmesis. Various surgical techniques had been described with variable success.

In this study, we compared the efficacy of Rotational Narrow Strip Conjunctival Graft with the conventional full conjunctival graft in pterygium excision. Patient will be follow up for a year after pterygium surgery. Outcome will be recurrence rate between the two groups at one year. Risk analysis of certain factors that affects the recurrence rate will be discussed.

ELIGIBILITY:
Inclusion Criteria:

1. Significant and symptomatic primary pterygium clinically requiring excision
2. Willingness to participate in research project and to attend research time

Exclusion Criteria:

1. Age < 21 years
2. Glaucoma in the study eye
3. Other concurrent ocular surface pathology
4. Infection of the ocular surface
5. Poor general health

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2007-07; Primary Completion 2008-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Recurrence Rate of Pterygium operated with Rotational Narrow Strip Conjunctival Graft and Full Conjunctival Graft Excision | 1 year

SECONDARY OUTCOMES:
Analysis of risk factors associated with recurrence of pterygium | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lo Sheau Kang, MBBS, Principal Investigator — University Malaya Eye Research Centre
Locations (1):
- Sarawak General Hospital, Kuching, Sarawak, Malaysia